CLINICAL TRIAL: NCT02380404
Title: Clinical Outcomes of a Cost-effective Implant Treatment in the Edentulous Upper Maxilla: Effectiveness of Removable Prosthesis Retained by 4 Implant-supported Locator-Attachments.
Brief Title: Effectiveness of Removable Prosthesis Retained by 4 Implant-supported Locator-Attachments
Acronym: LOC
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Université de Liège (Other); ITI International Team for Implantology, Switzerland (Other); Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Head of Clinic, University of Liege
Other Study IDs: 958_2013
Record Dates: First submitted 2014-03-06; First posted 2015-03-05 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Edentulous maxilla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Edentulous maxilla: Ibuprofen (600 mg - Film-coated Tablets) 3x/day before the surgery. Duration : 5 days Amoxicilline Teva (500 mg - dispersible tablets) 3x/day before the surgery. Duration : 16 days
  Interventions: Procedure: Implants-supported locators placement

INTERVENTIONS:
Procedure: Implants-supported locators placement — Antibiotics will be prescribed 1 day before surgery and continued for 5 days. Three calibrated surgeons will place 4 NN or RN Roxolid tissue level implants. Two implants have to be placed in the ANT region (lateral or canine) and 2 implants in the POST region (as distal as possible). Angulated implant and placement of implant in the tuberosity region can be considered.
  Other Names: Locators abutments; NN or RN Roxolid tissue level implants

SUMMARY:
1. Hypothesis/Specific aims

The aim of the present study proposal is to validate an implant treatment concept in the edentulous upper maxilla using four implants-supported locators abutments to retain removable prosthesis.

Specific aims:

* The primary objective of the study is to evaluate the implant and prosthodontics success rates of the proposed implant treatment approach after a follow-up period of 1, 3 and 5 years as well as the biological and prosthodontics complications.
* The secondary objective is to assess the evolution of patient centered outcomes with the suggested treatment in the maxilla. Oral health-related quality of life (OHRQoL) and patients' satisfaction relating to their prostheses will be considered.
* The third objective will be to compare the implant, prosthodontics and patient-centered outcomes according to the implant distribution; 4 anterior to maxillary sinus (ANT) versus 2 anterior implants and 2 implants in the maxillary tuberosity (POST).

Hypothesis:

* Implant survival rate using this treatment concept is similar to restoration with implant-supported fixed prosthesis, based on published data. No difference of implant survival rates is found between ANT and POST implant distribution.
* Prosthodontics survival rate using the following treatment concept is similar to the ones found with a bar, based on published data. The ANT implant distribution causes fewer prosthodontics complications compared to the POST implant distribution.
* There is a significant improvement in OHRQoL and patient satisfaction compared to the baseline OHRQoL observed with a conventional removable denture. The levels of improvement OHRQoL and patient satisfaction are similar for ANT and POST implant distributions.

DETAILED DESCRIPTION:
1.1 Background and significance

The effectiveness of mandibular overdentures retained by 2 dental implants and its impact on Oral Health-Related Quality of Life (OHRQoL) and patient satisfaction has been extensively documented over the last decades(1-6). According to recent systematic reviews, the implant survival rate of this oral rehabilitation concept reaches more than 95% (7-10). The scientific validation of the efficacy of such a rehabilitation concept has influenced the social security system of several countries like Belgium. Therefore, this treatment approach is nowadays considered as an evidence-based and cost-effective treatment option improving the function and quality of life of mandibular edentulous patients. Unfortunately, cost-effective treatment concept to restore the edentulous maxilla not has been widely documented (11). Many studies display high success rates of fixed implant-supported rehabilitations of the edentulous maxilla (12) but these treatment options remain costly and are therefore reserved to a limited social category of patients.

This work is important because there is a need to provide affordable and efficient implant treatment approaches to restore function and improve satisfaction and OHRQoL of patients with edentulous maxillae.

1.2 Preliminary studies in connection with new projects/continuing projects

Even though some authors have described implant survival rates of implant-retained overdentures in the upper maxilla (8, 13-16), most of the treatment approaches involves bars. The placement of 4 implants and individual attachments is a more cost-effective treatment modality that is poorly documented in the literature in terms of implants and prosthodontics outcomes but also on aspects assessing implant distribution, attachment types and improvement of patient centered outcomes. Therefore, further studies are needed to validate the placement of 4 implants and individual attachment as a reliable treatment modality.

1.3 Research design and methods

The study is designed as a single center prospective cohort study. The study protocol will be submitted to the Ethics Committee of the University Hospital of the University of Liège, Belgium.

A total of 30 patients with edentulous maxillae and at least one short span dentition (fixed) in the lower jaw will be included in the study.

The inclusion and exclusion criteria are listed below:

Inclusion criteria

* Physical status according to the American Society of Anesthesiologists (ASA) = 1, 2
* Wearing a complete upper denture that is adequate and in good conditions
* Signed informed consent form describing the purpose and process of the study

Exclusion criteria

* Uncontrolled periodontitis/peri-implantitis (lower jaw)
* Lack of bone for the placement of 4 implants of 3.3 diameter and 8 mm with bone regeneration.
* Tobacco use > 10cigarettes/day

Pre-treatment examination Clinical evaluation of the upper removable denture and the lower dentition will be done. Oral hygiene instructions will be given.

The patient fulfilling the inclusion criteria will be asked to complete 3 questionnaires for patient satisfaction and OHRQoL and socio-demographic conditions before explaining them the possibilities to be enrolled in a study in order to minimize the risk of bias.

The McGill Denture Satisfaction Instrument (17) will be used to evaluate patients' satisfaction relating to their prostheses. This questionnaire is a treatment-specific patient-based outcome assessing satisfaction relating to 6 aspects of the mandibular prosthesis: general satisfaction, comfort, stability, aesthetics, chewing ability (ease of chewing), chewing efficiency (ability to crush food in small particles), ease of cleaning, ability to speak and oral condition (condition of their mouth, which can refer to oral health status and was measured by "In general, are you satisfied with your oral condition?". The subjects will answer on 100 mm visual analogue scales (VAS) anchored by the words "not at all satisfied" and "extremely satisfied".

The Oral Health Impact Profile (OHIP-20) questionnaire will be used to assess oral health-related quality of life. This 20-item questionnaire measures self-reported impairment in edentulous populations within seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. The items will be rated on six-point Likert scales ("never" = 1, "rarely" = 2, "occasionally" = 3, "often" = 4, "very often" = 5 or "all of the time" = 6). OHIP-20s total range is therefore 20-120 points, lower scores indicating better oral health-related quality of life (4, 18, 19).

Data on gender, age, level of education, annual household revenue, marital status and lifestyle (living alone or with others) will be obtained from a standard socio-demographic questionnaire.

Cone beam CT s assessment After the informed consent is signed, a CT scan will be done and evaluated by 2 independent surgeons to potentially exclude some patients because of lack of bone availability. In case of disagreement, the case will be discussed.

Surgical procedures Once all patients have been enrolled in the study, the surgeries will be scheduled within the same week. Antibiotics will be prescribed 1 day before surgery and continued for 5 days. Three calibrated and confirmed surgeons will place 4 Narrow Neck (NN) or Regular Neck (RN) Roxolid tissue level implants (Institut Straumann, Basel Switzerland) according to the surgical protocol recommended by the manufacturer. The implant positions have to be determined previously at the time of CT scan evaluation by an agreement between the 2 operators and according to the bone availability. Two implants have to be placed in the lateral or canine region and 2 implants as distal as possible. The implants have to be placed with as parallels as possible. A maximum divergence of 10 will be tolerated. The flap design will be determined according to the available bone quantity and in order to emphasize an adequate quantity of keratinized tissue around the implants. A Cone Beam Computed Tomography (CBCT) scan will be done directly after surgery. Sutures will be performed with silk sutures and removed after 1 week. The removable (conventional) prostheses will be adapted to avoid any contact with the implants. Patients will be followed up at 4 and 8 weeks post-surgery, respectively. At 8 weeks, a panoramic x-ray will be done. If osseointegration is successful, the removable prostheses will be connected to the implants.

Prosthodontics procedures At 8 weeks, prosthesis will be connected to the implant with Locator . The type of Locator attachments will be chosen according to the implant angulation and soft tissue thickness. They will be torqued at 35 N/cm on the osseointegrated implants. Afterwards, the female connection will be fixed into the removable prosthesis with acrylic resin. The effectiveness of retention will be checked and the patient will be taught to put the denture in and out by himself. The occlusion will be controlled and adjusted after these manipulations if necessary.

Follow-up visits Patient will be followed at 1 week after Locator connections and then at 3, 6 and 12 months, respectively. Thereafter, patients were recalled annually. In case of any complications, the patient will be asked to directly contact one of the dentists responsible for the study.

Data collection Data will be collected into a remote and secured database. Automatic data check procedures will be implemented at data entry to warrant quality of the information stored. Access to the database will be limited to the study investigators and data will be kept confidential.

Statistical analyses Results will be summarized as mean and standard deviation (SD) for quantitative variables and as frequency tables for categorical findings at each time point. Longitudinal data will be displayed graphically and analyzed by the general linear mixed model which accounts for repeated values within patients. Success rates will be estimated and associated with 95% confidence intervals (95%CI). The significance level will be set at 5% (P<0.05). Data will be analyzed with Statistical Analyses Software (SAS and S-PLUS softwares).

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to ASA = 1, 2
* Wearing a complete upper denture that is adequate and in good conditions
* Signed informed consent form describing the purpose and process of the study

Exclusion Criteria:

* Uncontrolled periodontitis/peri-implantitis (lower jaw)
* Lack of bone for the placement of 4 implants of 3.3 diameter and 8 mm with bone regeneration.
* Tobacco use > 10cigarettes/day

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Department of Periodontology and Oral Surgery, CHU of Liège
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Implant outcomes | 5 years
  At each follow-up visit (3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years), a clinical exam including plaque assessment, bleeding on probing and mucosal palpation will be done. A CBCT scan will be done directly after surgery and at one year post-surgery. Specifically, the integration will be considered successful if the following parameters are met: (1) absence of recurring peri-implant infection with suppuration; (2) absence of persistent subjective complaints such as pain, foreign body sensation, and/or dysesthesia; (3) absence of a continuous radiolucency around the implant; and (4) absence of any detectable implant mobility. Marginal bone levels will be measured using CBCT radiograph at baseline and 1, 3 and 5 years follow-up, using the implant neck as reference point and calibrating them using Image J64. Marginal bone remodeling will be calculated accordingly. CBCT radiographs will be taken using the bisector technique.

SECONDARY OUTCOMES:
Prosthodontics success rates | 5 years
  At each follow-up visit (3 months, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years), the proper adaptation of the prosthesis, the retention of attachments and the mastication aptitude will be verified. A fracture of the Locator attachments will be considered as a prosthodontics failure and will directly influence the prosthodontics success rates. The possible prosthodontics complications, such as base fracture, attachment loss (unscrewing, or discementation) and loss of retention, will be recorded as prosthodontics complications and managed appropriately.

OTHER OUTCOMES:
Quality of life and self-assessment | 12 months
  The OHIP-20 and patient satisfaction questionnaires as described in the 'patient examination' section will be also submitted to the patients before at 3, 6 and 12 months after the connection of the removable prosthesis to the Locator attachments. Thereafter, the patients will receive these questionnaires annually.

CONTACTS AND LOCATIONS:
Overall Officials: France Lambert, Principal Investigator — CHU of Liège
Locations (2):
- Belgium (2):
  - Hospital University of Liège (CHU-Ulg), Liège
  - University Hospital of Liege, Liège

REFERENCES:
- [Background] Assuncao WG, Barao VA, Delben JA, Gomes EA, Tabata LF. A comparison of patient satisfaction between treatment with conventional complete dentures and overdentures in the elderly: a literature review. Gerodontology. 2010 Jun;27(2):154-62. doi: 10.1111/j.1741-2358.2009.00299.x. Epub 2009 May 6. PMID 19467020
- [Background] Awad MA, Locker D, Korner-Bitensky N, Feine JS. Measuring the effect of intra-oral implant rehabilitation on health-related quality of life in a randomized controlled clinical trial. J Dent Res. 2000 Sep;79(9):1659-63. doi: 10.1177/00220345000790090401. PMID 11023260
- [Background] Awad MA, Lund JP, Dufresne E, Feine JS. Comparing the efficacy of mandibular implant-retained overdentures and conventional dentures among middle-aged edentulous patients: satisfaction and functional assessment. Int J Prosthodont. 2003 Mar-Apr;16(2):117-22. PMID 12737240
- [Background] Awad MA, Rashid F, Feine JS; Overdenture Effectiveness Study Team Consortium. The effect of mandibular 2-implant overdentures on oral health-related quality of life: an international multicentre study. Clin Oral Implants Res. 2014 Jan;25(1):46-51. doi: 10.1111/clr.12205. Epub 2013 Jun 4. PMID 23735197
- [Background] Heydecke G, Penrod JR, Takanashi Y, Lund JP, Feine JS, Thomason JM. Cost-effectiveness of mandibular two-implant overdentures and conventional dentures in the edentulous elderly. J Dent Res. 2005 Sep;84(9):794-9. doi: 10.1177/154405910508400903. PMID 16109986
- [Background] Wismeijer D, Tawse-Smith A, Payne AG. Multicentre prospective evaluation of implant-assisted mandibular bilateral distal extension removable partial dentures: patient satisfaction. Clin Oral Implants Res. 2013 Jan;24(1):20-7. doi: 10.1111/j.1600-0501.2011.02367.x. Epub 2011 Nov 24. PMID 22111809
- [Background] Batenburg RH, Meijer HJ, Raghoebar GM, Vissink A. Treatment concept for mandibular overdentures supported by endosseous implants: a literature review. Int J Oral Maxillofac Implants. 1998 Jul-Aug;13(4):539-45. PMID 9714961
- [Background] Slot W, Raghoebar GM, Vissink A, Huddleston Slater JJ, Meijer HJ. A systematic review of implant-supported maxillary overdentures after a mean observation period of at least 1 year. J Clin Periodontol. 2010 Jan;37(1):98-110. doi: 10.1111/j.1600-051X.2009.01493.x. Epub 2009 Dec 7. PMID 19995402
- [Background] de Lange J, van Gool AV, Stoker G, Wismeijer D, van Waas R. An eight-year follow-up to a randomized clinical trial of aftercare and cost-analysis with three types of mandibular implant-retained overdentures. J Dent Res. 2007 Oct;86(10):920; author reply 920-1. doi: 10.1177/154405910708601003. No abstract available. PMID 17890666
- [Background] Stoker G, van Waas R, Wismeijer D. Long-term outcomes of three types of implant-supported mandibular overdentures in smokers. Clin Oral Implants Res. 2012 Aug;23(8):925-9. doi: 10.1111/j.1600-0501.2011.02237.x. Epub 2011 Jul 4. PMID 21722193
- [Background] Zembic A, Wismeijer D. Patient-reported outcomes of maxillary implant-supported overdentures compared with conventional dentures. Clin Oral Implants Res. 2014 Apr;25(4):441-50. doi: 10.1111/clr.12169. Epub 2013 Apr 15. PMID 23581398
- [Background] Lambert FE, Weber HP, Susarla SM, Belser UC, Gallucci GO. Descriptive analysis of implant and prosthodontic survival rates with fixed implant-supported rehabilitations in the edentulous maxilla. J Periodontol. 2009 Aug;80(8):1220-30. doi: 10.1902/jop.2009.090109. PMID 19656021
- [Background] Laurito D, Lamazza L, Spink MJ, De Biase A. Tissue-supported dental implant prosthesis (overdenture): the search for the ideal protocol. A literature review. Ann Stomatol (Roma). 2012 Jan;3(1):2-10. Epub 2012 May 3. PMID 22783448
- [Background] Slot W, Raghoebar GM, Vissink A, Meijer HJ. Maxillary overdentures supported by anteriorly or posteriorly placed implants opposed by a natural dentition in the mandible: a 1-year prospective case series study. Clin Implant Dent Relat Res. 2014 Feb;16(1):51-61. doi: 10.1111/j.1708-8208.2012.00459.x. Epub 2012 May 11. PMID 22577941
- [Background] Slot W, Raghoebar GM, Vissink A, Meijer HJ. A comparison between 4 and 6 implants in the maxillary posterior region to support an overdenture; 1-year results from a randomized controlled trial. Clin Oral Implants Res. 2014 May;25(5):560-6. doi: 10.1111/clr.12118. Epub 2013 Feb 13. PMID 23406268
- [Background] Michaud PL, de Grandmont P, Feine JS, Emami E. Measuring patient-based outcomes: is treatment satisfaction associated with oral health-related quality of life? J Dent. 2012 Aug;40(8):624-31. doi: 10.1016/j.jdent.2012.04.007. Epub 2012 Apr 20. PMID 22522414
- [Background] Allen F, Locker D. A modified short version of the oral health impact profile for assessing health-related quality of life in edentulous adults. Int J Prosthodont. 2002 Sep-Oct;15(5):446-50. PMID 12375458
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981